CLINICAL TRIAL: NCT01893528
Title: Study to Assess the Safety and Tolerability of Ascending Single Doses of REGN2009 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: R2009-HV-1304
Record Dates: First submitted 2013-06-21; First posted 2013-07-09 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- REGN2009 dose level 1 (Experimental): Cohort A - REGN2009 or placebo; Cohort B - Patients on existing (non-exclusionary) medications + (REGN2009 or placebo)
  Interventions: Drug: REGN2009; Other: placebo
- REGN2009 dose level 2 (Experimental): Cohort C - REGN2009 or placebo; Cohort D - Patients on existing (non-exclusionary) medications + (REGN2009 or placebo)
  Interventions: Drug: REGN2009; Other: placebo
- REGN2009 dose level 3 (Experimental): Cohort E - REGN2009 or placebo; Cohort F - Patients on existing (non-exclusionary) medications + (REGN2009 or placebo)
  Interventions: Drug: REGN2009; Other: placebo

INTERVENTIONS:
Drug: REGN2009
Other: placebo

SUMMARY:
This is a phase 1, randomized, double-blind, placebo-controlled first-in-human (FIH) study to assess the safety and tolerability of ascending single doses of REGN2009 administered to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women ages 18 to 65 years inclusive
2. Body mass index between 18.0 kg/m^2 and 30.0 kg/m^2, inclusive

Exclusion Criteria:

1. Pregnant or breast-feeding women
2. Any clinically significant abnormalities observed during screening (day -21 to day -2)
3. Known history of human immunodeficiency virus (HIV) antibody; and/or positive hepatitis B surface antigen, and/or positive hepatitis C antibody at the screening visit
4. History of drug or alcohol abuse within a year prior to the screening visit (day -21 to day -2)
5. Hospitalization for any reason within 60 days of the screening visit (day -21 to day -2)
6. Participation in any clinical research study within 30 days of the screening visit (day -21 to day -2) or within 5 half-lives of the investigational drug or therapy being studied (whichever is longer)
7. History of a hypersensitivity reaction to doxycycline or similar compound
8. Any medical or psychiatric condition which, in the opinion of the investigator, would place the subject at risk, interfere with participation in the study or interfere with the interpretation of the study results
9. Previous adverse experience to any biological investigational or therapeutic agent
10. Sexually active men or women of childbearing potential who are unwilling to practice adequate contraception during the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial and not all inclusion/ exclusion criteria are listed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Number of TEAEs | day 1 to day 106/ visit 15
  The primary endpoint in this study is the incidence and severity of Treatment Emergent Adverse Events (TEAEs) in healthy volunteers treated with REGN2009 or placebo reported from day 1 (baseline) to the completion of the study on day 106/ visit 15.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- United States (2):
  - Baltimore, Maryland
  - Cincinnati, Ohio